CLINICAL TRIAL: NCT01895959
Title: Quantifications of Biochemical Changes of Synovial Fluid and Cartilage Matrix in Osteoarthritic Knee After Hyaluronic Acid Injection Using Novel MRI (Magnetic Resonance Imaging) and NMR (Nuclear Magnetic Resonance) Techniques
Brief Title: To Look at the Characteristics of Synovial Fluid and Cartilage Matrix in Osteoarthritic Knee After Hyaluronic Acid Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Ferring-Euflexxa
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis (OA); hyaluronic acid injection
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Euflexxa (Other): EUFLEXXA® is a hyaluronate hydrogel produced from bacteria, in a phosphate-buffered saline solution. It is given as a three week treatment regimen. It involves injecting of 2cc or 20mg intra-articularly once per week.
  Interventions: Drug: Euflexxa; Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: Euflexxa — Euflexxa will be injected weekly for 3 consecutive weeks on the knee joint.
  Other Names: hyaluronic acid injection
Device: Magnetic Resonance Imaging (MRI) — MRI of the knee will be acquired during baseline (a week prior to the treatment), follow up visit 1 (1 week after treatment) and follow up visit 2 (3 months after treatment).

SUMMARY:
The purpose of this study is to identify novel imaging markers for characterizing the biochemical profiles in synovial fluid and cartilage matrix in OA knee joints after intra-articular HA (Euflexxa) injection using high field NMR and MRI techniques.

We hypothesize that:

1. High-field HRMAS NMR spectroscopy will provide sensitive measures for biochemical changes within knee synovial fluid after HA injection;
2. Baseline HRMAS spectroscopy, in particular N-acetyl peaks, as well as early changes of glutamate will predict patient response of pain relief after HA injection;
3. MR cartilage T1p and T2 quantifications will provide sensitive measures for biochemical changes within knee cartilage matrix after HA injection. Specifically cartilage T1p and T2 will decrease in patients who respond to the treatment, indicating potential beneficial effects of HA injection to cartilage preservation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* Symptomatic knee OA as defined by the American College of Rheumatology criteria
* Kellgren-Lawrence grade I, II or III on prior x-rays (take within 6 months of screening visit)
* knee pain score >40 mm on a 100 mm visual analogue scale for > 15 days in the last month
* NSAIDs permitted if the dose has been stable for at least one month prior to baseline and stays stable during the study
* Have been recommended for Euflexxa treatment by physician
* Knee effusion based on clinical exam or imaging

Exclusion Criteria:

* Any contraindication to MRI (pregnancy, metallic fragments in the eyes, vascular clips, Pacemakers etc)
* History of knee replacement
* Known sensitivity or allergy to any component of Euflexxa
* Inflammatory arthritis
* Previously received viscosupplementation therapy within 6 months of study enrollment
* Intra-articular injection of corticosteroid to study joint within the past 3 months
* Arthroscopic or open surgery within the previous 12 months or planned surgery to the study joint
* Concomitant medications of oral/parenteral corticosteroids
* Morbid obesity defined as body mass index (BMI) >40 kg/m2
* Active malignancy; an active systemic infection; recent high impact or high energy trauma (clinically defined) to the study joint
* Large knee effusion based on clinical exam or imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojuan Li, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF - China Basin Imaging Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Subjects treated with Euflexxa
Period: Overall Study
Arm/Group | Treatment
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.17 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: To Identify Imaging Markers for Characterizing the Biochemical Profiles in Synovial Fluid and Cartilage in Knee OA After HA Injection
Description: The study will demonstrate the feasibility of using MRI and NMR techniques to quantify biochemical changes in synovial fluid and cartilage matrix in OA knees after HA injection.
Time Frame: 3 months
Population: The PI left institution and all efforts to locate outcome measure data have been exhausted and therefore cannot be reported.
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: To Quantify Synovial Fluid Biochemical Changes Using High Field HRMAS NMR Spectroscopy
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: To Quantify Cartilage Matrix Changes Using MR T1p ad T2 Mapping at 3T MRI
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=12)
knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes